CLINICAL TRIAL: NCT01799031
Title: Reducing Work Disability in Breast Cancer Survivors
Brief Title: Educational Intervention for Reducing Work Disability in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OS12115; NCI-2012-03055 (Registry Identifier: NCI Trial ID); 2012-0729 (Other: Institutional Review Board); A536130 (Other: UW Madison); SMPH\ORTHOPEDIC&REHAB\PT (Other: UW Madison)
Record Dates: First submitted 2013-02-21; First posted 2013-02-26 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer; Cancer Survivor
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (WISE) (Experimental): Patients receive access to the WISE web-based educational intervention to help BCS manage their symptoms, identify ergonomic workplace problems and risks, and implement ergonomic modifications. Patients also receive standard of care comprising symptom management therapies and a pamphlet on employment rights.
  Interventions: Other: internet-based intervention; Procedure: management of therapy complications; Other: educational intervention; Other: questionnaire administration; Procedure: quality-of-life assessment
- Arm II (control) (Active Comparator): Patients receive standard of care comprising symptom management therapies and a pamphlet on employment rights.
  Interventions: Procedure: management of therapy complications; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: internet-based intervention — Receive access to the WISE web-based educational intervention
  Arms: Arm I (WISE)
Procedure: management of therapy complications — Receive standard of care
  Other Names: complications of therapy, management of
Other: educational intervention — Receive access to the WISE web-based educational intervention
  Other Names: intervention, educational
  Arms: Arm I (WISE)
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This randomized clinical trial studies an educational intervention for reducing work disability in breast cancer survivors. Web sites providing symptom management education may be an effective method to help breast cancer survivors reduce work disability after treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility and usability of the Work Ability Improvement Through Symptom Management and Ergonomic Strategies (WISE) and empirically evaluate its effect on short-term work ability among breast cancer survivors (BCS).

SECONDARY OBJECTIVES:

I. Explore individual and workplace factors associated with work ability in BCS.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive access to the WISE web-based educational intervention to help BCS manage their symptoms, identify ergonomic workplace problems and risks, and implement ergonomic modifications. Patients also receive standard of care comprising symptom management therapies and a pamphlet on employment rights.

ARM II: Patients receive standard of care comprising symptom management therapies and a pamphlet on employment rights.

After completion of study treatment, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer
* Employed at time of cancer diagnosis (defined as paid employment > 20 hours/week)
* Within six months of completion of active treatment
* Working during treatment or intending to return to work following active treatment
* Computer and internet access

Exclusion Criteria:

* Patients who do not intend to continue/resume working following treatment
* Develop distant metastases or progressive disease
* Prior diagnosis of malignancy at any other site except for in situ carcinomas of the cervix or non-melanomatous skin cancers

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Usability of the WISE website as assessed by responses to a 5-point Likert scale | 3 months
  The primary analysis of the effect of the WISE intervention on work ability will be performed using a Wilcoxon rank sum test.
Usability of the WISE website as assessed by responses to a 5-point Likert scale | 6 months
  The primary analysis of the effect of the WISE intervention on work ability will be performed using a Wilcoxon rank sum test.
Work ability, assessed by the Work Limitations Questionnaire (WLQ) | Baseline
Work ability, assessed by the WLQ | 3 months
Work ability, assessed by the WLQ | 6 months
Individual factors, including symptoms assessed using the Symptom Bother-Revised scale (SB-R) and MD Anderson Symptom Inventory (MDASI), socio-demographic factors, individual disease factors, and treatment factors | Baseline
Individual factors, including symptoms assessed using the SB-R and MDASI, socio-demographic factors, individual disease factors, and treatment factors | 3 months
Individual factors, including symptoms assessed using the SB-R and MDASI, socio-demographic factors, individual disease factors, and treatment factors | 6 months
Workplace factors, including work history, job characteristics, job control, job support, and level of job stress using the Job Content Questionnaire (JCQ) | Baseline
Workplace factors, including work history, job characteristics, job control, job support, and level of job stress using the JCQ | 3 months
Workplace factors, including work history, job characteristics, job control, job support, and level of job stress using the JCQ | 6 months

SECONDARY OUTCOMES:
Feasibility measures, including participation/dropout rates, patient satisfaction, usability/satisfaction with WISE, knowledge/use of self-care symptom management/ergonomic strategies, and use of ergonomic/symptom management strategies, and barriers | Up to 6 months
Self-car symptom management strategies used (if any), workplace strategies implemented, and barriers to implementation | Up to 6 months
Individuals self-reported work ability, using the Work Ability Index (WAI) | Up to 6 months
Employment status | Up to 6 months
Change in job performance or difficulty performing work tasks | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sesto, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/